CLINICAL TRIAL: NCT01210963
Title: Central Corneal Thickness After Overnight IOP Monitoring With SENSIMED Triggerfish
Brief Title: Central Corneal Thickness With SENSIMED Triggerfish
Acronym: 09/08
Status: Completed | Type: Observational
Sponsor: Sensimed AG (Industry)
Responsible Party: Priv. Doz. Dr. med. Thomas Klink, Universitätsklinikum Würzburg, Augen- und Poliklinik
Other Study IDs: 09/08
Record Dates: First submitted 2010-09-27; First posted 2010-09-29 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-03

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SENSIMED Triggerfish
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish — Contact lens-based Sensor with recording system for continuous monitoring of IOP fluctuation

SUMMARY:
Investigation of the occurrence of possible corneal swelling after continuous Intraocular pressure (IOP) monitoring with a contact lens-based Sensor during the sleeping period.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma and ocular hypertension scheduled for overnight hospitalisation
* stable IOP-lowering treatment since at least 4 weeks before study
* at least 18 years
* having provided informed consent

Exclusion Criteria:

* contact lens wear within the last 2 years
* contraindication for silicone lean wear
* corneal abnormality in either eye
* ocular infection or inflammation
* history of ocular surgery within the last 3 months
* full-frame metal glasses during IOP monitoring with SENSIMED Triggerfish
* pregnancy and lactation
* patients not able to understand the nature of the research
* patients under tutelage
* patients committed to an institution by virtue of an order issued either by the courts or by an authority
* simultaneous participation in other clinical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma and ocular hypertension patients, at least 18 years old and with stable IOP-lowering treatment (if any).
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Pachymetry (central corneal thickness) | after 8 hours nocturnal continuous IOP monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Klink, PD Dr. med, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- Augen- und Poliklinik, Universitätsklinikum Würzburg, Würzburg, Germany